CLINICAL TRIAL: NCT06306885
Title: Effects of Early Sleep After Action Observation and Motor Imagery in Patients Undergoing Immobilization After Surgery for Metacarpal and Phalangeal Fractures
Brief Title: Effects of Early Sleep After Action Observation and Motor Imagery After Metacarpal Fracture Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF23/03
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Hand Injuries; Action Observation; Motor Imagery
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AOMI-sleep (Experimental): Observation and imagination of video-clips with motor contents before sleeping
  Interventions: Behavioral: Action observation plus motor imagery followed by sleep
- AOMI-control (Active Comparator): Observation and imagination of video-clips with motor contents in the morning
  Interventions: Behavioral: Action observation plus motor imagery
- Control (Sham Comparator): Observation and imagination of landscapes video-clips
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Action observation plus motor imagery followed by sleep — Participants will be asked to observe video-clips showing motor contents immediately before sleeping
  Arms: AOMI-sleep
Behavioral: Action observation plus motor imagery — Participants will be asked to observe video-clips showing motor contents at least 12 hours before sleeping
  Arms: AOMI-control
Behavioral: Control — Participants will be asked to observe video-clips showing landscapes before sleeping
  Arms: Control

SUMMARY:
The study aimed to investigate the effects of early sleep after action observation and motor imagery (AOMI) training sessions on manual dexterity in patients with hand immobilization after surgical fixation for metacarpals and phalanges fractures.

Fifty-one patients with hand immobilization for surgical fixation of IV or V metacarpals or first phalanges fractures will be randomized into AOMI-sleep (n=17), AOMI-control (n=17), and Control (n=17) group. AOMI-sleep and AOMI-control groups will perform an AOMI-training before sleeping or in the morning respectively, while Control group will be asked to observe landscape video-clips. Participants will be assessed for manual dexterity, hand range of motion, hand disability and quality of life at baseline before and after the training and at 1 month after the training end.

DETAILED DESCRIPTION:
The study aimed to investigate the effects of early sleep after action observation and motor imagery (AOMI) training sessions on manual dexterity in patients with hand immobilization after surgical fixation for metacarpals and phalanges fractures.

Fifty-one patients with right hand immobilization for surgical fixation of IV or V metacarpals or first phalanges fractures will be randomized into an AOMI-sleep (n=17), AOMI-control (n=17), and Control (n=17) group. AOMI-sleep and AOMI-control groups will perform a 2-week AOMI-training including transitive manual dexterity tasks between 8:00 and 10:00 p.m. or between 8:00 and 10:00 a.m. respectively, while Control group participants will be asked to observe landscape video-clips between 8:00 and 10:00 p.m. Participants will be assessed for manual dexterity (Purdue Pegboard Test and kinematic indexes during Nine Hole Peg Test), hand range of motion (Total Active Motion) hand disability (Quick-DASH) and quality of life (EQ5D) at baseline (1 week after surgery), training end (3 weeks after surgery) and 1 month after the training end (7 weeks after surgery).

ELIGIBILITY:
Inclusion Criteria:

* Surgical fixation for IV or V MTC or P1 fracture at the level of the right hand
* Age 18-40 years old
* Right-hand dominance

Exclusion Criteria:

* Damage to additional hand structure requiring surgery (e.g. tendons, ligaments and nerves)
* Occurrence of left upper limb injuries
* Post-surgical complications (e.g. CPRS)
* Immobilization <12 or >30 days
* Diagnosis of neurological/musculoskeletal conditions
* Sports or activities requiring advanced manual skills or sleep deprivation
* History of psychiatric disorders
* Sleep disorders (e.g. insomnia, OSAS, REN or Non-REM behavioural disorders)
* Medication affecting the physiological sleep pattern

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Purdue Pegboard Test | Before and after 2 weeks of training and at 1 month follow-up
  Manual dexterity test

SECONDARY OUTCOMES:
Changes in kinematic indexes during Nine Hole Peg Test | Before and after 2 weeks of training and at 1 month follow-up
  Manual dexterity test with kinematic indexes recording
Changes in Visual Analogue Scale | Before and after 2 weeks of training and at 1 month follow-up
  Scale assessing perceived pain
Changes in Quick-DASH | Before and after 2 weeks of training and at 1 month follow-up
  Questionnaire assessing upper limb disability
Changes in EQ5D | Before and after 2 weeks of training and at 1 month follow-up
  Questionnaire assessing quality of life
Changes in Total Active Motion | Before and after 2 weeks of training and at 1 month follow-up
  Measurement of the range of motion of V and IV fingers
Hand-grip strength | 1-month follow-up
  Test of maximal strength with a dynamometer

IPD SHARING:
Plan to Share IPD: No